CLINICAL TRIAL: NCT07255547
Title: Arthrosocpic Treatment of Knee Chondral Lesions: Clinical, MRI and Histologic Comparison Between the Use of PRP vs ADSCs in Addition to Marrow Stimulation Techniques
Brief Title: PRP vs AD-SVF in Addition to Marrow Stimulation for Knee Chondral Lesion
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi dell'Aquila (Other)
Collaborators: Arthrex GmbH (Industry)
Responsible Party: Principal Investigator, Andrea Vespasiani, MD, Università degli Studi dell'Aquila
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23/2019; EMEA-18060 (Other Grant/Funding Number: Arthrex GmbH)
Record Dates: First submitted 2025-08-27; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-08

CONDITIONS: Knee Chondral Lesion
Keywords: PRP; AD-SVF; knee arthroscopy; cartilage; adipose tissue; microfracture; stromal vascular fraction
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PRP (Active Comparator): In this arm, patients undergo arthroscopic microfracture of the chondral lesion and PRP injection.
  Interventions: Procedure: Bone Marrow Stimulation; Drug: PRP injection
- PRP + AD-SVF (Experimental): In this arm, patients undergo arthroscopic microfracture of the chondral lesion and PRP and AD-SVF injection.
  Interventions: Procedure: Bone Marrow Stimulation; Combination Product: stromal vascular fraction (SVF)

INTERVENTIONS:
Procedure: Bone Marrow Stimulation — All patients underwent an arthroscopic procedure (that further confirmed the preoperative diagnosis; i.e. monocompartmental chondral lesion - Outerbridge grade IV) including a concomitant bone marrow stimulation technique (microfracture). According to the technique described by Steadman, the cartilaginous lesion underwent preliminary debridement to remove the damaged cartilage and form a stable edge of healthy tissue and subsequent microfracture with an arthroscopic pick to stimulate the subchondral unit regenerative response.
  Other Names: knee arthroscopy; Steadman microfracture
Combination Product: stromal vascular fraction (SVF) — After bone marrow stimulation technique, patients were randomly assigned to one of the two treatment arms (allocation ratio 1:1). 40 patients underwent PRP injection while the other 40 underwent PRP + AD-SVF injections.
  Other Names: PRP injection
  Arms: PRP + AD-SVF
Drug: PRP injection — After bone marrow stimulation technique, patients were randomly assigned to one of the two treatment arms (allocation ratio 1:1). 40 patients underwent PRP injection while the other 40 underwent PRP + AD-SVF injections.
  Arms: PRP

SUMMARY:
The goal of this clinical trial is to learn if PRP and adipose-derived stem cells (AD-SVF) enhance healing after knee microfracture for chondral lesions. It will also learn about the safety of the procedure. The main questions it aims to answer are:

Do PRP and AD-SVF get better results than PRP alone in patients undergoing arthroscopic microfracture for knee monocompartmental cartilage injuries? What medical problems do participants have when taking drug ABC? Researchers will compare PRP + AD-SVF to PRP alone to see if PRP + AD-SVF work better to treat knee cartilage injuries.

Participants will:

Undergo knee microfracture and biologics injections at the end of the arthroscopic procedure (PRP+AD-SVF vs PRP).

Visit the clinic for checkups and tests at baseline and at 3, 6, 12 months post-treatment, and then annually.

ELIGIBILITY:
Inclusion Criteria:

* knee pain and functional limitation for at least three months, monocompartmental chondral lesion < 2 cm2, age over 18, and BMI between 18.5 and 30

Exclusion Criteria:

* previous major surgery on the same knee, concomitant chondral lesions in other knee compartments, being diagnosed with knee or hip osteoarthritis, knee instability, flexion deficit > 20° or extension deficit >15°, genu valgum or genu varum > 20°, patients with Hb values < 11 g/dL or platelet < 150000/µL, patients in therapy with antiaggregants or anticoagulants or immunosuppressive agents, pregnancy, and the following comorbidities: hematological/neurologic/metabolic/rheumatic diseases, neoplastic disorders or history of local infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in knee clinical function questionnaire (KOOS) | From preoperatively (baseline) until the end of the study, up to 60 months.
  Knee Injury Osteoarthritis Outcome Score is a self-administered questionnaire and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. The resulting scores are then transformed to a scale from 0 to 100, with 0 representing extreme knee problems and 100 representing no knee problems. The scores on this scale represent the percentage of the total possible score that the person achieved.

SECONDARY OUTCOMES:
Knee pain assessment | From preoperatively (baseline) until the end of the study, up to 60 months.
  Pain intensity was measured using the Visual Analogue Scale (VAS).
Adverse events after the procedure | Until the end of the study, up to 60 months.
  Adverse events such as knee swelling and pain with longer recovery time
Other Patient-Reported Outcome Measures | From preoperatively (baseline) to the end of the study, up to 60 months.
  Overall physical and mental health-related quality of life was assessed with the 12-item Short Form Survey (SF-12). The SF-12 was constructed using questions drawn from each of the 8 dimensions of the MOS 36 item Short Form Survey (SF-36). It is designed to have similar performance to the SF-36, while taking less time to complete.Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12).
  Additionally, the IKDC questionnaire was used to measure knee symptoms, functional limitations, and sports activity. An ordinal scoring system is used to assign a score of 0 to responses that signify the lowest level of function or the highest level of symptoms for each item. The IKDC Subjective Knee Evaluation Form is graded by adding the results of each item's scores, and then converting the result to a 0-100 scale. Higher scores indicate higher levels of function and lower levels of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- San Salvatore Hospital, L’Aquila, Abruzzo, Italy

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication

REFERENCES:
- [Background] Bora P, Majumdar AS. Adipose tissue-derived stromal vascular fraction in regenerative medicine: a brief review on biology and translation. Stem Cell Res Ther. 2017 Jun 15;8(1):145. doi: 10.1186/s13287-017-0598-y. PMID 28619097
- [Background] Prodromidis AD, Charalambous CP, Moran E, Venkatesh R, Pandit H. The role of Platelet-Rich Plasma (PRP) intraarticular injections in restoring articular cartilage of osteoarthritic knees. A systematic review and meta-analysis. Osteoarthr Cartil Open. 2022 Nov 5;4(4):100318. doi: 10.1016/j.ocarto.2022.100318. eCollection 2022 Dec. PMID 36474791
- [Background] Srinivasan V, Ethiraj P, Agarawal S, H S A, Parmanantham M. Comparison of Various Modalities in the Treatment of Early Knee Osteoarthritis: An Unsolved Controversy. Cureus. 2023 Jan 11;15(1):e33630. doi: 10.7759/cureus.33630. eCollection 2023 Jan. PMID 36788843
- [Background] Cong B, Sun T, Zhao Y, Chen M. Current and Novel Therapeutics for Articular Cartilage Repair and Regeneration. Ther Clin Risk Manag. 2023 Jun 20;19:485-502. doi: 10.2147/TCRM.S410277. eCollection 2023. PMID 37360195
- [Background] Welton KL, Logterman S, Bartley JH, Vidal AF, McCarty EC. Knee Cartilage Repair and Restoration: Common Problems and Solutions. Clin Sports Med. 2018 Apr;37(2):307-330. doi: 10.1016/j.csm.2017.12.008. PMID 29525030
- [Background] Mirza MZ, Swenson RD, Lynch SA. Knee cartilage defect: marrow stimulating techniques. Curr Rev Musculoskelet Med. 2015 Dec;8(4):451-6. doi: 10.1007/s12178-015-9303-x. PMID 26411978

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT07255547/Prot_SAP_ICF_000.pdf